CLINICAL TRIAL: NCT03244488
Title: Cholinergic Correlates of Impaired Cognitive Ability in HIV-Associated Neurocognitive Disorders
Brief Title: Mental Ability Challenge Study in Adults With and Without HIV
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Asante Kamkwalala, Graduate Research Assistant, Vanderbilt University Medical Center
Other Study IDs: 150929
Record Dates: First submitted 2017-07-27; First posted 2017-08-09 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: HIV-1-infection; Aging, Premature; Cognitive Impairment; Memory Impairment; HIV-Associated Cognitive Motor Complex
MeSH Terms: conditions — Aging, Premature; Cognitive Dysfunction; Memory Disorders; AIDS Dementia Complex | interventions — Mecamylamine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples collected from all participants for routine screening labs and APOE genotyping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV-Positive: Patients will be administered each of 4 possible treatments: high dose (5 mcg/kg) scopolamine, high dose (20 mg) mecamylamine, a low dose combination (2.5mcg/kg and 10 mg) of scopolamine and mecamylamine, or placebo.
  Interventions: Drug: Scopolamine Injectable Product; Drug: Mecamylamine Pill
- HIV-Negative: Patients will be administered each of 4 possible treatments: high dose (5 mcg/kg) scopolamine, high dose (20 mg) mecamylamine, a low dose combination (2.5mcg/kg and 10 mg) of scopolamine and mecamylamine, or placebo.
  Interventions: Drug: Scopolamine Injectable Product; Drug: Mecamylamine Pill

INTERVENTIONS:
Drug: Scopolamine Injectable Product — 2.5 or 5 mcg/kg of scopolamine via IV
Drug: Mecamylamine Pill — 10 or 20mg of mecamylamine orally

SUMMARY:
It is estimated that by 2016, nearly 50% of HIV-positive individuals in the US will be aged 50 or older, and up to 60% of those will experience some degree of cognitive impairment as they age. The purpose of this study is to evaluate the contribution of the neuronal cholinergic receptor system to the cognitive impairments seen in adults aging with chronic HIV Infection. By using anti-cholinergic challenge drugs to reversibly "stress" cognitive functioning, the investigators hope to understand whether the presence of the HIV virus in the brain impairs the neural system necessary for normal cognition, more than would be expected from normal cognitive aging.

DETAILED DESCRIPTION:
This study is intended to evaluate the involvement of the neuronal cholinergic receptor system in the accelerated cognitive aging profile seen in adults living with chronic HIV-1 infection. It is estimated by the CDC that by the year 2016, nearly 50% of the US' HIV-positive population will be 50 or older. The HIV-1 virus is known to enter the CNS very rapidly after initial infection, and cause a pattern of persistent neural inflammation, which is deleterious to neurons and glia. This damage is believed to be the basis of cognitive impairment associated with long-term chronic HIV infection, known as HIV-Associated Neurocognitive Disorders (HAND). Successful introduction of Anti-Retroviral Treatment (ART) has greatly reduced the likelihood of progressing to the most severe category of HAND (HIV-Associated Dementia), however the mild and moderate forms (Asymptomatic Neurocognitive Impairment and Mild Neurocognitive Disorder, respectively) are still fairly common even in adults declared "virally suppressed", with little to no detectable peripheral viral DNA/RNA. Prior studies have shown that over the lifetime, more than 50% of adults diagnosed with HIV will experience some degree of cognitive impairment as they age. Some of these changes may be due to cholinergic dysfunction. The acetylcholinergic receptor system is necessary for normal cognitive performance, and is active during working memory, executive functioning, attention, and learning tasks. It has been shown that as the human brain ages, cognitive ability begins to decline, and correlates with declining acetylcholinergic activity. The cholinergic theory of cognitive aging postulates that this loss of activity at cholinergic receptors with age is at least partly responsible for poorer cognitive performance in aging. I will use this model to examine the impact of HIV infection on cholinergic system functioning. This study will use a well-established anti-cholinergic drug challenge model to evaluate cognitive performance in domains of cognitive functioning relevant to cholinergic functioning. Under conditions of temporary muscarinic or nicotinic blockade, or a combination of both, I aim to explore the contribution of putative cholinergic receptor dysfunction to the observed symptoms of HAND. I also intend to determine whether age and HIV-status interact to produce an accelerated pattern of cholinergic cognitive aging that would indicate that older adults with HIV are at higher risk for more rapid cognitive aging than HIV-negative individuals. If successful, the outcome of this study would support the future exploration of novel pro-cholinergic medications to treat cognitive symptoms of HAND, which may improve quality of life for adults living with chronic HIV infection, as they survive into old age.

ELIGIBILITY:
Inclusion Criteria:

1. 35 years of age or older;
2. HIV-Positive (must be on ART's for at least 6 months, most recent viral load (within 6 months) <50, CD4+ count >200, must be diagnosed HIV-positive at least 5 years) or HIV-Negative, At-Risk Individuals
3. Able and willing to give written informed consent
4. Negative urine pregnancy test
5. Adequate visual and auditory acuity to allow neuropsychological testing.

Exclusion Criteria:

1. Unmanaged HIV Infection, identified by no current medication regimen or the presence of one or more AIDS-defining conditions
2. Fagerstrom cigarettes per day (CPD) score of '2' indicating heavy use of nicotine
3. An ART regimen including a Protease Inhibitor Medication
4. A documented history of cardiac disease or abnormal ECG at Screening
5. Current alcohol or substance abuse, particularly intravenously
6. Current use of psychoactive medications (antipsychotics, benzodiazepines, etc.)
7. Current Axis I or Axis II psychiatric disorder
8. History of myocardial infarction in the past year or unstable or severe cardiovascular disease

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-Positive Healthy older adults and HIV-Negative Healthy older adults
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Cognitive Outcome - Lower verbal memory score | 2 hours
  Cognitive performance will be more significantly impaired by study medications in HIV-positive participants relative to HIV-negative participants, indicating impairment of cholinergic neurotransmitter system.

SECONDARY OUTCOMES:
Age and HIV-Status Interaction - Slower CRTreaction time | 2 hours
  Older age and positive HIV status will interact to more significantly impair cognitive performance as measured by reaction time on the Choice Reaction Time task under the influence of study medications, than either variable alone.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No